CLINICAL TRIAL: NCT05162898
Title: Henan Cancer Hospital, Affiliated Cancer Hospital of Zhengzhou University
Brief Title: Radiofrequency Ablation Combined With Toripalimab and Lenvatinib in the Treatment of Short-term Recurrent Hepatocellular Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-245
Record Dates: First submitted 2021-11-28; First posted 2021-12-17 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Hepatocellular Cancer
Keywords: PD-1 Inhibitor; Radiofrequency ablation; toripalimab; lenvatinib; Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — toripalimab; lenvatinib; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GROUP 1 (Experimental)
  Interventions: Drug: toripalimab; Drug: Lenvatinib; Device: Radiofrequency ablation

INTERVENTIONS:
Drug: toripalimab — 240mg,ivgtt, every three weeks as a cycle, the first day of each cycle.
Drug: Lenvatinib — 12mg (weight ≥60kg) or 8mg (weight <60kg) orally, once a day
Device: Radiofrequency ablation — ultrasound-guided percutaneous radiofrequency ablation of recurrent hepatocellular carcinoma

SUMMARY:
This study is a multi-center, prospective, single-arm, open-design phase II clinical study, mainly to explore the clinical effectiveness and safety of radiofrequency ablation combined with anti-PD-1 antibody toripalimab and lenvatinib in patients with short-term recurrence of hepatocellular carcinoma.

DETAILED DESCRIPTION:
Primary endpoint: Recurrence-free survival time (RFS). Secondary endpoints: safety (incidence of adverse events); time to recurrence (TTR); time to local recurrence (TTLR); 12-month recurrence-free survival rate; overall survival (OS); 12 months and 24 Month overall survival rate.

Treatment plan: Patients undergo radiofrequency ablation, 3-5 days after radiofrequency ablation, lenvatinib 12 mg (body weight ≥ 60 kg) or 8 mg (body weight <60 kg) orally, once a day; toripalimab is a fixed dose of 240 mg, once every 3 weeks, intravenous infusion on the first day of each cycle, the infusion time is no less than 60 minutes.Combination therapy until tumor recurrence, disease progression, death or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, ≤75 years old, no gender limit;
2. Primary hepatocellular carcinoma confirmed pathologically and clinically;
3. After radical resection and 2 months after radiofrequency ablation, no tumor lesions were found in imaging examination (MRI, CT plain scan enhancement), and recurrence and no metastasis of liver cancer occurred within 1 year after surgery;
4. ECOG score 0-1 points (Appendix 1);
5. Recurrent liver cancer meets Milan criteria: single tumor diameter ≤ 5 cm or multiple tumors less than 3 with maximum diameter ≤ 3 cm, no large vessel infiltration, no lymph node or extrahepatic metastasis;
6. Child-Pugh liver function classification: A, B;
7. Expected survival> 6 months;
8. Sufficient organ function: ①No growth factor and blood component support is required within 2 weeks before enrollment; ②Heart function: no heart disease or coronary heart disease, the patient's heart function is grade 1-2; ③Within 7 days before enrollment , Has sufficient liver and kidney function, suitable laboratory indicators (untreated): HGB≧9.0g/dl, neutrophils≧1,500/mm3, PLT≧50x109/L, serum ALB≧28g/L, TBIL< 2 mg/dL, ALT, AST<5 times the upper limit of normal value, Bun, Cr<1.5 times the upper limit of normal value, INR<1.7 or prolonged PT<3s;
9. Patients with normal blood pressure or hypertension should use antihypertensive drugs to control their blood pressure within the normal range;
10. The fasting blood sugar of diabetic patients should be controlled at ≤8mmol/L through hypoglycemic drugs;
11. No other serious diseases that conflict with this plan (such as autoimmune diseases, immunodeficiency, organ transplantation);
12. No history of other malignant tumors;
13. Women of childbearing age must have a negative blood pregnancy test within 7 days, and subjects of childbearing age must use appropriate contraceptive measures during the test and within 6 months after the test;
14. The patient himself agrees to participate in this clinical study and signs the "Informed Consent".

Exclusion Criteria:

1. Previously received radiotherapy, chemotherapy, hormone therapy or molecular targeted therapy;
2. Patients with distant metastasis confirmed by imaging;
3. The subject has previously or simultaneously suffered from other malignant tumors (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
4. The subjects who have been treated with toripalimab or other PD-1/PD-L1 treatments in the past cannot be included in the group; the subject is known to have been allergic to macromolecular protein preparations, or is known to be allergic to any of the components of teriprizumab;
5. The subject has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis , Nephritis, hyperthyroidism, reduced thyroid function; subjects suffering from vitiligo or asthma in childhood has been completely relieved, and can be included in adults without any intervention; subjects requiring bronchodilators for medical intervention can not be included;
6. The subject is using immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve immunosuppressive purposes (dose>10mg/day prednisone or other curative hormones), and within 2 weeks before enrollment Still in use;
7. Cardiac clinical symptoms or diseases that are not well controlled, such as: (1) Heart failure above NYHA level 2 (2) Unstable angina (3) Myocardial infarction occurred within 1 year (4) Supraventricular with clinical significance Or patients with ventricular arrhythmia in need of treatment or intervention;
8. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg>2g/L), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy;
9. The patient currently (within 3 months) has gastrointestinal diseases such as esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension, or active bleeding from unresected tumors, or the investigator determines Other conditions that may cause gastrointestinal bleeding and perforation;
10. Past or current severe bleeding (bleeding >30 ml within 3 months), hemoptysis (>5 ml fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient cerebral deficiencies) within 12 months Blood attack);
11. Past and current patients with objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc.;
12. Subjects with congenital or acquired immune deficiencies, such as HIV infection, or active hepatitis (transaminase does not meet the selection criteria, hepatitis B reference: HBV DNA ≥10⁴/ml; hepatitis C reference: HCV RNA ≥103/ml); chronic Carriers of hepatitis B virus, HBV DNA <2000 IU/ml (<104 copies/ml), must receive antiviral therapy at the same time during the trial period before they can be included in the group;
13. The subject is participating in other clinical studies or is less than one month away from the end of the previous clinical study; the subject may receive other systemic anti-tumor treatments during the study period;
14. The subject is known to have a history of psychotropic drug abuse, alcohol abuse or drug abuse;
15. Re-examination within 2 months after the operation, the patient with tumor recurrence or metastasis confirmed by imaging examination.
16. The investigator believes that it should be excluded from this study. For example, according to the investigator's judgment, the subject has other factors that may cause the study to be terminated halfway, such as other serious diseases (including mental illness) that require combined treatment. Serious laboratory examination abnormalities, accompanied by family or social factors, will affect the safety of subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
RFS | up to 36 months
  Recurrence-free survival time

SECONDARY OUTCOMES:
safety | 24 months
  Adverse event rate
TTR | up to 36 months
  time to recurrence
1-year RFS% | 12 months
  1-year recurrence-free survival rate
OS | 2025
  overall survival
1-year OS% | 12 months
  1-year overall survival rate
2-year OS% | 24 months
  2-year overall survival rate

IPD SHARING:
Plan to Share IPD: No